CLINICAL TRIAL: NCT04462835
Title: Feasibility, Effectiveness and Safety of 3000 Hysteroscopies in Outpatient Setting
Brief Title: Feasibility, Effectiveness and Safety of Outpatient Hysteroscopy
Acronym: FESHA
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-FES-2019-96
Record Dates: First submitted 2020-07-06; First posted 2020-07-08 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Hysteroscopy; Outpatient
Keywords: Hysteroscopy; outpatient; Gold standard

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study Objective: The main objective of the study is to assess the feasibility, effectiveness and safety of outpatient hysteroscopies performed in our Office Hysteroscopy Unit.

Design: Retrospective observational study of prospectively collected data from the Office Hysteroscopy Unit database.

Setting: Tertiary care university hospital

Patients: Three thousand patients who consecutively attended an ambulatory hysteroscopy in our centre from may 2008 to october 2019

Interventions: The Office hysteroscopy was performed with several rigid 5-6 mm diameter devices when indicated with a diagnostic and/or therapeutic purpose

DETAILED DESCRIPTION:
Retrospective observational study of our prospectively collected database of 3000 consecutive hysteroscopies performed from may 2008 to october 2019 in our Office Hysteroscopy Unit (OHU).

All the patients who attended an ambulatory hysteroscopy in our centre during the study period were included. There were not any exclusion criteria and all data were prospectively collected in a computer database.

The primary endpoint was to determine the main results of the Outpatient Hysteroscopy Unit in terms of feasibility, effectiveness and safety. Feasibility was defined as the proportion of explorations that could be satisfactorily performed. Effectiveness was evaluated through the percentage of cases that were solved in our outpatient setting and did not require the operating room to complete their diagnosis or treatment. Safety was assessed as the percentage of complications registered.

In addition, we registered the intensity of the pain perceived by the patient with a Verbal Numerical Rating Scale (VNRS) (from 0 to 10) during the procedure and ten minutes later.

All the hysteroscopies were performed in our Office Hysteroscopy Unit by three experienced gynaecologists who performed the hysteroscopy assisted by a nurse.

For pain and anxiety management, a painkiller (ibuprofen 600 mg) and an anxiolytic (diazepam 5 mg) were orally dispensed to all patients 30 minutes before the procedure. Cervical preparation with Misoprostol (400 mcg, intravaginal administration 4-6 hours before the test) was administered only in cases of anticipated or previous failed cervical passage. Paracervical anaesthesia was administered in selected cases of several pain during the passage through the cervical canal. Premenopausal women were asked to take desogestrel 75 mg, at least 30 days prior to the procedure for endometrial preparation and if the patient was unwilling to take the medication, the procedure was preferably performed in the early follicular phase.

Hysteroscopy was performed with the several diagnostic and therapeutic rigid devices available in our Office Hysteroscopy Unit in 5-6 mm diameter: mechanical instruments (scissors and forceps), bipolar electrode (Versapoint ®), bipolar Gubini resector (Colibrí®) and mechanical morcelators (Myosure® and Truclear®), They have been set up gradually in our Unit. Saline solution 0.9% was used as a distention media with an automated pressure delivery system and he vaginoscopic approach was performed.

ELIGIBILITY:
Inclusion Criteria:

* All the patients who attended an ambulatory hysteroscopy in our centre.

Exclusion Criteria:

* There were not any exclusion criteria.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who attended an ambulatory hysteroscopy in our centre.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Feasibility: proportion of hysteroscopies that could be satisfactorily performed | 3 months
  Feasibility refers to the proportion of hysteroscopies that could be satisfactorily performed
Efectiveness: Percentage of cases that were solved in our outpatient setting and did not require the operating room to complete their diagnosis or treatment | 3 months
  Percentage of cases that were solved in our outpatient setting and did not require the operating room to complete their diagnosis or treatment
Safety: Percentage of complications registered | 3 months
  Percentage of complications registered.

SECONDARY OUTCOMES:
Pain during the hysteroscopy and 10 minutes later: Verbal Numerical Rating Scale (VNRS) | 3 months
  The intensity of the pain perceived by the patient with a Verbal Numerical Rating Scale (VNRS) (from 0 which is no pain to 10 which is the worst pain ever imagined) during the procedure and ten minutes later.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Simo Gonzalez, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Background] Bakour SH, Jones SE, O'Donovan P. Ambulatory hysteroscopy: evidence-based guide to diagnosis and therapy. Best Pract Res Clin Obstet Gynaecol. 2006 Dec;20(6):953-75. doi: 10.1016/j.bpobgyn.2006.06.004. Epub 2006 Nov 20. PMID 17116420
- [Background] Capmas P, Pourcelot AG, Giral E, Fedida D, Fernandez H. Office hysteroscopy: A report of 2402 cases. J Gynecol Obstet Biol Reprod (Paris). 2016 May;45(5):445-50. doi: 10.1016/j.jgyn.2016.02.007. Epub 2016 Apr 4. PMID 27055773
- [Background] Bennett A, Lepage C, Thavorn K, Fergusson D, Murnaghan O, Coyle D, Singh SS. Effectiveness of Outpatient Versus Operating Room Hysteroscopy for the Diagnosis and Treatment of Uterine Conditions: A Systematic Review and Meta-Analysis. J Obstet Gynaecol Can. 2019 Jul;41(7):930-941. doi: 10.1016/j.jogc.2018.10.002. Epub 2018 Dec 7. PMID 30528838
- [Background] Krins T. Outpatient hysteroscopy. Aust N Z J Obstet Gynaecol. 2017 Oct;57(5):E10. doi: 10.1111/ajo.12662. No abstract available. PMID 28967691
- [Background] Diwakar L, Roberts TE, Cooper NA, Middleton L, Jowett S, Daniels J, Smith P, Clark TJ; OPT trial collaborative group. An economic evaluation of outpatient versus inpatient polyp treatment for abnormal uterine bleeding. BJOG. 2016 Mar;123(4):625-31. doi: 10.1111/1471-0528.13434. Epub 2015 May 25. PMID 26011792
- [Background] Campo R, Santangelo F, Gordts S, Di Cesare C, Van Kerrebroeck H, De Angelis MC, Di Spiezio Sardo A. Outpatient hysteroscopy. Facts Views Vis Obgyn. 2018 Sep;10(3):115-122. PMID 31191845